CLINICAL TRIAL: NCT06432751
Title: Pre-operative Exposure to SGLT2 Inhibitors and Post-operative Acute Renal Failure in Cardiac Surgery
Acronym: SGLT2i-PO-AKI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0517
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury; Cardiac Surgery; Sodium/Glucose Cotransporter Inhibitor 2
Keywords: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Adults patients with pre-operative simplified predictive risk index for renal replacement therapy after cardiac surgery ≥2, with cardiac surgery performed in Louis Pradel Hospital between 08/2022 and 02/2024.
  Interventions: Other: Post Operative Acute Kidney Injury

INTERVENTIONS:
Other: Post Operative Acute Kidney Injury — Serum creatinine increase by 0.3 mg/dl within 48 h OR Serum creatinine ≥ 1.5-1.9 times baseline within 7 days
  Baseline creatinine is defined as the last pre-operative value available in the medical file

SUMMARY:
Cardiac surgery with cardiopulmonary bypass exposes patients to the risk of post-operative acute kidney injury. In the specific setting of cardiac surgery, acute kidney injury is often of multifactorial origindue to particular haemodynamic mechanisms, renal hypoxia, or damage linked in the inflammatory reaction or haemolysis.

In recent years, inhibitors of the sodium/glucose co-transporter type 2 have demonstrated their relevance in reducing the morbidity and mortality associated with chronic or acute heart failure and chronic kidney disease. These drugs were initially developed to optimise glycaemic control in diabetic patients. They are currently recommended as part of the management of diabetic patients at high cardiovascular risk, patients with systolic and/or diastolic heart failure, and patients with chronic kidney disease.

Some pharmacodynamic properties of SGLT2i suggest that they could have a beneficial effect in preventing the onset of acute kidney injury, but also that they could lead to potentially deleterious effects in renal haemodynamic in specific situations.

The aim of the study was to estimate the impact of pre-operative exposure to SGLT2i on the occurrence of post-operative acute kidney injury in high-risk renal patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Cardiac surgery with cardiopulmonary bypass
* Presenting a simplified renal risk score ≥ 2 points defined as follows:

  * Pre-operative glomerular filtration rate (≤ 60; ≤ 30 mL/min/1.73m2): 1-2 points
  * Diabetes requiring treatment: 1 point
  * LVEF ≤ 40%: 1 point
  * Previous cardiac surgery: 1 point
  * Pre-operative intra-aortic counter pulsation: 1 point
  * Non elective surgery: 1 point
  * Surgery other than closure of an atrial septal defect or coronary bypass surgery: 1 point

Exclusion Criteria:

* Haemodialysis prior to surgery
* Acute kidney injury prior to surgery as defined in the primary endpoint. If this criterion is not available, patients will only be included if glomerular filtration rate estimated by the CKD-EPI formula is ≥75 mL/min/1.73m2.
* Death in the operating theatre
* Opposition of the patient to the use of his/her health data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1200 patients admitted in the Louis Pradel Hospital for cardiac surgery in the study period
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Post-operative acute kidney injury | Baseline creatinine is defined as the last pre-operative value available in the medical file Variation of the creatinine was explored in the first 7 postoperative days
  Serum creatinine increase by 0.3 mg/dl within 48 h
Post-operative acute kidney injury | Baseline creatinine is defined as the last pre-operative value available in the medical file Variation of the creatinine was explored in the first 7 postoperative days
  Serum creatinine ≥ 1.5-1.9 times baseline within 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital cardiologique Louis Pradel Groupe Hospitalier Est, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No